CLINICAL TRIAL: NCT01116947
Title: Fosrenol for Enhancing Dietary Protein Intake in Hypoalbuminemic Dialysis Patients (FrEDI) Study: An Investigator Initiated Study
Brief Title: Fosrenol for Enhancing Dietary Protein Intake in Hypoalbuminemic Dialysis Patients (FrEDI) Study
Acronym: FrEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: DaVita, Inc. (Industry); Shire (Industry)
Responsible Party: Principal Investigator, kamyar kalantar-zadeh, md phd mph, Professor of medicine, pediatrics and epidemiology, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LABioMed 13892-01
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: End-Stage Renal Disease
Keywords: Hypoalbuminemia; Hyperphosphatemia; Phosphorus; Protein; CKD; Dialysis; Meals; Lanthanum; End-Stage Renal Disease (ESRD); Dietary Protein Intake (DPI); Dietary Phosphorus Binding (DPB); Protein-Energy Wasting (PEW); Sources of Dietary Phosphorus
MeSH Terms: conditions — Kidney Failure, Chronic; Hypoalbuminemia; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Active Comparator): 1. Treatment Arm (CASES) will receive high protein meals during thrice weekly hemodialysis in-center (each meal includes ~50 g of protein, ~850 Cal, and phos/protein ratio <10 mg/g) PLUS dietary counseling to continue similar high protein intake with low phosphorus to protein ratio and to avoid foods with high preservative content. Fosrenol 1.0 to 1.5 g per meal will be prescribed (use of pill crusher will be recommended) and will be titrated based on bi-weekly phosphorus levels.
  Interventions: Other: Meals during hemodialysis accompanied by lanthanum carbonate to control phosphorus
- Control Arm (CONTROLS) (Active Comparator): 2. Control Arm (CONTROLS) will receive salad boxes in-center (no protein, low calorie) and routine dietary counseling and will continue pre-existing phosphorus binder regimen.
  Interventions: Other: Meals during hemodialysis accompanied by lanthanum carbonate to control phosphorus

INTERVENTIONS:
Other: Meals during hemodialysis accompanied by lanthanum carbonate to control phosphorus — Based on the hypothesis that the efficacy and potency of Fosrenol enables increasing dietary protein intake and provision of meals during dialysis treatment for improving nutritional status in malnourished dialysis patients with a low serum albumin (<4.0 g/dL) while serum phosphorus can be effectively controlled with the target range of 3.5 to 5.5 mg/dL

SUMMARY:
Protein-energy wasting, as reflected by a serum albumin <4.0 g/dL, is very common in maintenance hemodialysis (MHD) patients and associated with poor clinical outcomes including high death rates. Hyperphosphatemia, reflected by serum phosphorus level >5.5 mg/dL, is also common disorder and associated with increased death risk in the same population. The traditional dietary intervention to control hyperphosphatemia is to restrict protein intake. This, however, may worsen protein-energy wasting as recently showed in large epidemiologic data, which indicated that the best survival was observed in MHD patients with increased protein intake while serum phosphorus could be controlled. We hypothesize that the provision of high protein diet will be possible if a potent phosphorus binder (Fosreonl™) will be prescribed simultaneously. Hence, we propose to conduct a randomized controlled trial in 110 hypoalbuminemic (albumin <4.0 mg/dL) MHD patients in several DaVita dialysis facilities in Los Angeles South Bay area. After 1:1 randomization, we will provide the participating subjects (the INTERVENTION group) with 8 weeks of high protein meals in form of prepared meal boxes (50 g protein, 850 Cal, and a phosphorus to protein ratio of <10 mg/gm) during each hemodialysis treatment, along with 0.5 to 1.5 g Fosrenol, to be titrated if necessary; as well as dietary counselling to maintain a high dietary protein intake at home (with same or similar binder regimen) for 8 weeks and to avoid food items with high phosphorus based additives. Meals will be prepared at Harbor-UCLA GCRC Bio-nutrition Department. We have reviewed and tested the feasibility of meal preparation and distribution system and the related logistics. The CONTROL group will also receive meal boxes but the meal contains low Calorie (<50 Cal) and almost zero protein (<1 g) diet (such as salads) during each hemodialysis treatment. These patients will continue their pre-existing phosphorus control regimens. As outcome variables, we will examine change in serum albumin over the 8 weeks of intervention. We will also examine changes in dietary protein and serum phosphorus in the 2 groups after 8 weeks of intervention. Quality of life and patient satisfaction will also be examined before and towards the end of the intervention phase. Given our ongoing 2-year study with a similar operation known as the AIONID Study and given DaVita dieticians'' collaboration and support, we anticipate successful recruitment, retention and data analyses within 8 to 12 months.

DETAILED DESCRIPTION:
RATIONALE:

Based on the hypothesis that the efficacy and potency of Fosrenol enables increasing dietary protein intake and provision of meals during dialysis treatment for improving nutritional status in malnourished dialysis patients with a low serum albumin (<4.0 g/dL) while serum phosphorus can be effectively controlled with the target range of 3.5 to 5.5 mg/dL.

STUDY PROCEDURE:

1. In all subjects: Recommend adequate dietary protein intake to achieve or maintain an nPCR (nPNA) above 1.0 g/kg/day for 2 months. Encourage aggressive increase in protein intake while avoiding high phos/protein ratio esp. higher intake of egg whites, meat, fish, poultries, legumes, etc. via counseling by renal dietician (RD) and/or study staff.
2. Both groups will receive free meal boxes during the first 60 min of HD treatment for 8 weeks (24 meals during 24 HD treatment sessions). Cases will receive high protein meals (~50 gm, with phos/protein ratio <10 mg//gm), whereas controls will receive salad with almost no protein.
3. In CASES (n=55): Switch binder simultaneously to (or start) Fosrenol 500 mg to 1,500 per meal/snack, according to the meal size at different times of the day. Recommend crushing the pills using the pill-crusher that will be provided to subjects, and recommend placing or sprinkling Fosrenol pieces on the food. Titrate the dose every 2 weeks according to serum phosphorus.
4. In CONTROLLS (n=55): Continue the same binder (other than Fosrenol). In All subjects: Titrate the binder as indicated to control serum phosphorus <5.5 mg/dL.

SAFETY ENDPOINTS:

1. Routine safety measures for food ingestion and binder administration
2. Bi-weekly measures of minerals and monthly measures of PTH

STATISTICAL METHODS:

The t test, the chi square test, and the Mann-Whitney rank sum test to compare the baseline characteristics of intervention and control participants in serum albumin and other measures. To simplify presentation of results, some Likert scale responses will be dichotomized. The corresponding P values will be based on the complete ordinal scales used by participants to respond to questions quality of life, satisfaction, and food intake and about how often they eat meals from specific fast-food restaurants.

ELIGIBILITY:
Inclusion Criteria:

1. Prevalent hypoalbuminemic hemodialysis patients with a serum albumin <4.0 g/dL and capable of oral food intake
2. Adult (18-85 years) hemodialysis patients for 3 months or longer, capable of eating food independently
3. Protein energy wasting as evident by serum albumin <4.0 g/dL
4. Not receiving Fosrenol for the past 2 weeks

   Exclusion Criteria:
5. Not willing to sign the written consent form
6. Any condition that can interfere with increasing dietary protein intake, e.g. inability to eat or to maintain ingested food (OK to be on vitamin D agents including paricalcitol, calcitriol, doxercalciferol, ergocalciferol and cholecalciferol; or cinacalcet)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
1. Change in serum albumin by +0.2 g/dl or higher over 2 months, i.e., from baseline (Month 0) to Month 2 (main outcome measure) | 2 months

SECONDARY OUTCOMES:
2. Percentage of serum phosphorus between 3.5 and 5.5 mg/dL | 2 months
3. Change in nPCR (nPNA) by +0.1 g/kg/day | 2 months
4. Change in protein intake via food frequency questionnaire x 2 (baseline vs. after 2 months) | 2 months
5. Change in post-dialysis dry weight | 2 months
6. Changes in calcium, PTH, and alkaline phosphatase | 2 months
7. Patients satisfaction and quality of life (KDQOL36) | 2 months
8. RD and MD satisfaction per questionnaires | 2 months
9. Change in other nutritional or inflammatory markers (CRP, TIBC, MIS, SGA) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamyar Kalantar-Zadeh, MD, MPH, PhD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Background] Kovesdy CP, Anderson JE, Kalantar-Zadeh K. Outcomes associated with serum phosphorus level in males with non-dialysis dependent chronic kidney disease. Clin Nephrol. 2010 Apr;73(4):268-75. doi: 10.5414/cnp73268. PMID 20353734
- [Background] Noori N, Kalantar-Zadeh K, Kovesdy CP, Bross R, Benner D, Kopple JD. Association of dietary phosphorus intake and phosphorus to protein ratio with mortality in hemodialysis patients. Clin J Am Soc Nephrol. 2010 Apr;5(4):683-92. doi: 10.2215/CJN.08601209. Epub 2010 Feb 25. PMID 20185606
- [Background] Kalantar-Zadeh K, Gutekunst L, Mehrotra R, Kovesdy CP, Bross R, Shinaberger CS, Noori N, Hirschberg R, Benner D, Nissenson AR, Kopple JD. Understanding sources of dietary phosphorus in the treatment of patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 Mar;5(3):519-30. doi: 10.2215/CJN.06080809. Epub 2010 Jan 21. PMID 20093346
- [Background] Shinaberger CS, Greenland S, Kopple JD, Van Wyck D, Mehrotra R, Kovesdy CP, Kalantar-Zadeh K. Is controlling phosphorus by decreasing dietary protein intake beneficial or harmful in persons with chronic kidney disease? Am J Clin Nutr. 2008 Dec;88(6):1511-8. doi: 10.3945/ajcn.2008.26665. PMID 19064510
- [Background] Noori N, Sims JJ, Kopple JD, Shah A, Colman S, Shinaberger CS, Bross R, Mehrotra R, Kovesdy CP, Kalantar-Zadeh K. Organic and inorganic dietary phosphorus and its management in chronic kidney disease. Iran J Kidney Dis. 2010 Apr;4(2):89-100. PMID 20404416
- [Background] Kovesdy CP, Kalantar-Zadeh K. Bone and mineral disorders in pre-dialysis CKD. Int Urol Nephrol. 2008;40(2):427-40. doi: 10.1007/s11255-008-9346-7. PMID 18368510
- [Background] Kalantar-Zadeh K, Kuwae N, Regidor DL, Kovesdy CP, Kilpatrick RD, Shinaberger CS, McAllister CJ, Budoff MJ, Salusky IB, Kopple JD. Survival predictability of time-varying indicators of bone disease in maintenance hemodialysis patients. Kidney Int. 2006 Aug;70(4):771-80. doi: 10.1038/sj.ki.5001514. Epub 2006 Jul 5. PMID 16820797
- [Background] Shinaberger CS, Kilpatrick RD, Regidor DL, McAllister CJ, Greenland S, Kopple JD, Kalantar-Zadeh K. Longitudinal associations between dietary protein intake and survival in hemodialysis patients. Am J Kidney Dis. 2006 Jul;48(1):37-49. doi: 10.1053/j.ajkd.2006.03.049. PMID 16797385
- [Background] Mehrotra R, Martin KJ, Fishbane S, Sprague SM, Zeig S, Anger M; Fosrenol Overview Research Evaluation Study for Early Experience Study Group. Higher strength lanthanum carbonate provides serum phosphorus control with a low tablet burden and is preferred by patients and physicians: a multicenter study. Clin J Am Soc Nephrol. 2008 Sep;3(5):1437-45. doi: 10.2215/CJN.04741107. Epub 2008 Jun 25. PMID 18579668